CLINICAL TRIAL: NCT06428981
Title: (Holistic Health Care) Influence of Surgical Intervention on the Body-mind-spirit of Patients Undergoing Cervical Spine Surgery
Brief Title: Surgical Intervention on the Body-mind-spirit of Patients With Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202200381B0
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2022-04

CONDITIONS: Cervical Spine Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spine surgery (Other): The inclusion criteria consisted of patients over the age of 20 who were diagnosed with degenerative cervical diseases, including herniation of the intervertebral disc, ossification of the posterior longitudinal ligament, and spinal stenosis, resulting in cervical radiculopathy, or degenerative cervical myelopathy, and were scheduled to undergo anterior discectomy with fusion surgery.
  Interventions: Other: degenerative cervical diseases

INTERVENTIONS:
Other: degenerative cervical diseases — Including herniation of the intervertebral disc, ossification of the posterior longitudinal ligament, and spinal stenosis, resulting in cervical radiculopathy, or degenerative cervical myelopathy, and were scheduled to undergo anterior discectomy with fusion surgery.

SUMMARY:
The study aimed to evaluate if surgical intervention in patients with degenerative cervical diseases improves quality of life (QOL), lowers pain-induced mental impairment, improves psychologic health, and promotes spiritual well-being.

DETAILED DESCRIPTION:
Degenerative cervical disease induces cervical radiculopathy and myelopathy, which have a significant impact on the patients' health. The study aimed to evaluate if surgical intervention in patients with degenerative cervical diseases improves quality of life (QOL), lowers pain-induced mental impairment, improves psychologic health, and promotes spiritual well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 20 who were diagnosed with degenerative cervical diseases, including herniation of the intervertebral disc, ossification of the posterior longitudinal ligament, and spinal stenosis, resulting in cervical radiculopathy, or degenerative cervical myelopathy, and were scheduled to undergo anterior discectomy with fusion surgery.

Exclusion Criteria:

* Patients who were unable to attend follow-up visits or complete the questionnaires, and those patients who expressed doubts or were unable to provide satisfactory responses regarding the trial.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Quality of life, mental health, pain relief, and spiritual health before surgery | Before surgery
  The outcomes were assessed using the 36-item Short Form Health Survey Quality of Life Scale (SF-36) before surgery.
Quality of life, mental health, pain relief, and spiritual health before surgery | Before surgery
  The outcomes were assessed using the Patient Health Questionnaire-9 (PHQ9) scale before surgery.
Quality of life, mental health, pain relief, and spiritual health before surgery | Before surgery
  The outcomes were assessed using the Pain Disability Questionnaire (PDQ) scale before surgery.
Quality of life, mental health, pain relief, and spiritual health before surgery | Before surgery
  The outcomes were assessed using the Holistic Well-being Scale (HWS) scale before surgery.
Quality of life, mental health, pain relief, and spiritual health after surgery | six months after surgery
  The outcomes were assessed using the 36-item Short Form Health Survey Quality of Life Scale (SF-36) six months after surgery.
Quality of life, mental health, pain relief, and spiritual health after surgery | six months after surgery
  The outcomes were assessed using the Patient Health Questionnaire-9 (PHQ9) scale six months after surgery.
Quality of life, mental health, pain relief, and spiritual health after surgery | six months after surgery
  The outcomes were assessed using the Pain Disability Questionnaire (PDQ) scale six months after surgery.
Quality of life, mental health, pain relief, and spiritual health after surgery | six months after surgery
  The outcomes were assessed using the Holistic Well-being Scale (HWS) scale six months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan